CLINICAL TRIAL: NCT06282107
Title: Effectiveness and Safety of Bilateral Superselective Adrenal Arterial Embolization (BiSAAE) for Resistant Hypertension
Brief Title: Effectiveness and Safety of BiSAAE for Resistant Hypertension.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiSAAE-RHT
Record Dates: First submitted 2024-02-18; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral superselective adrenal arterial embolization (Experimental): Selectively injects 1.5-2.5 mL ethanol into bilateral adrenal artery to ablate part of the adrenal gland; irbesartanhydrochlorothiazide 162.5 mg/d, amlodipine 5 mg/d
  Interventions: Procedure: BiSAAE
- traditional triple antihypertensive treatment (Active Comparator): irbesartanhydrochlorothiazide 162.5 mg/d, amlodipine 5 mg/d
  Interventions: Procedure: traditional triple antihypertensive treatment

INTERVENTIONS:
Procedure: BiSAAE — SAAE is a catheter-based percutaneous transluminal procedure which selectively injects ethanol into bilateral adrenal artery to ablate part of the adrenal gland for suppression of excessive aldosterone and catecholamines
  Arms: Bilateral superselective adrenal arterial embolization
Procedure: traditional triple antihypertensive treatment — traditional triple antihypertensive treatment
  Arms: traditional triple antihypertensive treatment

SUMMARY:
Hypertension is a common problem, affecting >1.1 billion people worldwide. Unfortunately, fewer than one in five treated patients with hypertension have their blood pressure (BP) under control. The increasing number of people with uncontrolled BP despite the use of three or more antihypertensive agents at optimal or maximally tolerated doses, with one of those agents preferably being a diuretic has been described as the resistant hypertension (RH). Achieving BP control is essential because patients with hypertension who have uncontrolled BP have significantly higher rates of all-cause, cardiovascular, heart disease and cerebrovascular disease mortality compared to normotensive individuals, whereas mortality risk in patients with well-controlled BP does not differ from that in normotensive individuals. There are a number of potential factors that contribute to the suboptimal control of hypertension, including medication non-adherence and prescribing inertia. This highlights the limitations of purely pharmacological approaches for the effective management of hypertension. In fact, the activation of the renin-angiotensin-aldosterone system (RAAS) and sympatho-adrenomedullary system play a pathogenic role in triggering and sustaining RH. Superselective adrenal arterial embolization (SAAE) is a catheter-based percutaneous transluminal procedure which selectively injects ethanol into adrenal artery to ablate part of the adrenal gland for suppression of excessive aldosterone and catecholamines. Over the last decade, unilateral SAAE has emerged as a potential treatment option for patients with primary aldosteronism. Whether this approach can be extrapolated to patients with RH is unclear. We thus set out to perform a randomized trial to compare the safety and efficacy of bilateral SAAE with antihypertensive medications in treating RH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 30-65 years old.
* Patients with resist hypertension (office systolic blood pressure ≥140 mmHg, and/or office diastolic blood pressure ≥90 mmHg, and/or 24-h average systolic blood pressure ≥130 mmHg) with rational lifestyle change and triple antihypertensive drugs (irbesartanhydrochlorothiazide 162.5 mg/d, amlodipine 5 mg/d) for at least 4 weeks.
* Informed consent signed and agreed to participate in this trial.

Exclusion Criteria:

* Secondary hypertension
* Adrenergic insufficiency.
* adrenocortical insufficiency
* Renal failure eGFR<60 mL/min/1.73 m2
* Heart failure with NYHA grade Ⅱ-Ⅳ grade or unstable angina, severe cardiovascular and cerebrovascular stenosis, myocardial infarction, intracranial aneurysm, stroke and other acute cardiovascular events.
* Acute infections, tumors and severe arrhythmias, psychiatric disorders, drugs or alcohol addicts.
* Liver dysfunction or the following history of liver disease: AST or ALT 3 times higher than the upper limit, liver cirrhosis, history of hepatic encephalopathy, esophageal variceal history or portal shunt history.
* Fertile woman without contraceptives.
* Coagulation dysfunction.
* Pregnant women or lactating women.
* Participated in other clinical trials or admitted with other research drugs within 3 months prior to the trial.
* Any surgical or medical condition which can significantly alter the absorption, distribution, metabolism, or excretion of any study drug.
* Allergy or any contraindications for the study drugs, contrast agents and alcohol.

History of depression, schizophrenia or vascular dementia.

-Refused to sign informed consent

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of 24-h average systolic blood pressure | 6-month
  Difference in the change of 24-h average systolic blood pressure between the intervention and control group
Change of 24-h average systolic blood pressure | 12-month
  Difference in the change of 24-h average systolic blood pressure between the intervention and control group
Change of 24-h average systolic blood pressure | 3-month
  Difference in the change of 24-h average systolic blood pressure between the intervention and control group

SECONDARY OUTCOMES:
Change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure | 6-month
  Difference in the change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure between the intervention and control group
Change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure | 3-month
  Difference in the change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure between the intervention and control group
Change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure | 12-month
  Difference in the change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure between the intervention and control group
Change of home systolic and diastolic pressure | 6-month
  Difference in the change of home systolic and diastolic pressure between the intervention and control group
Change of home systolic and diastolic pressure | 12-month
  Difference in the change of home systolic and diastolic pressure between the intervention and control group
Change of home systolic and diastolic pressure | 3-month
  Difference in the change of home systolic and diastolic pressure between the intervention and control group
Difference in the change of office systolic and diastolic pressure between the intervention and control group | 6-month
  Difference in the change of office systolic and diastolic pressure between the intervention and control group
Difference in the change of office systolic and diastolic pressure between the intervention and control group | 12-month
  Difference in the change of office systolic and diastolic pressure between the intervention and control group
Difference in the change of office systolic and diastolic pressure between the intervention and control group | 3-month
  Difference in the change of office systolic and diastolic pressure between the intervention and control group
Difference in the change of blood electrolytes (K+, Na + in mmol/L) between the intervention and control group | 6-month
  Difference in the change of blood electrolytes (K+, Na + in mmol/L) between the intervention and control group
Difference in the change of blood electrolytes (K+, Na + in mmol/L) between the intervention and control group | 12-month
  Difference in the change of blood electrolytes (K+, Na + in mmol/L) between the intervention and control group
Difference in the change of blood electrolytes (K+, Na + in mmol/L) between the intervention and control group | 3-month
  Difference in the change of blood electrolytes (K+, Na + in mmol/L) between the intervention and control group
Change of plasma aldosterone | 6-month
  Difference in the change of plasma aldosterone (pg/mL) between the intervention and control group
Change of plasma aldosterone | 12-month
  Difference in the change of plasma aldosterone (pg/mL) between the intervention and control group
Change of plasma aldosterone | 3-month
  Difference in the change of plasma aldosterone (pg/mL) between the intervention and control group
Change of plasma cortisol | 6-month
  Change of plasma cortisol
Change of plasma cortisol | 12-month
  Change of plasma cortisol
Change of plasma cortisol | 3-month
  Change of plasma cortisol
Change of plasma renin measured | 6-month
  Difference in the change of plasma renin (pg/ml) between the intervention and control group
Change of plasma renin measured | 12-month
  Difference in the change of plasma renin (pg/ml) between the intervention and control group
Change of plasma renin measured | 3-month
  Difference in the change of plasma renin (pg/ml) between the intervention and control group
Change of liver enzymes | 6-month
  Difference in the change of liver enzymes (ALT, AST in IU/L) between the intervention and control group
Change of liver enzymes | 12-month
  Difference in the change of liver enzymes (ALT, AST in IU/L) between the intervention and control group
Change of liver enzymes | 3-month
  Difference in the change of liver enzymes (ALT, AST in IU/L) between the intervention and control group
Change of kidney function | 6-month
  Difference in the change of serum creatinine in umol/L between the intervention and control group
Change of kidney function | 12-month
  Difference in the change of serum creatinine in umol/L between the intervention and control group
Change of kidney function | 3-month
  Difference in the change of serum creatinine in umol/L between the intervention and control group
Change of fasting blood glucose | 6-month
  Difference in the change of fasting blood glucose in mmol/L between the intervention and control group
Change of fasting blood glucose | 3-month
  Difference in the change of fasting blood glucose in mmol/L between the intervention and control group
Change of fasting blood glucose | 12-month
  Difference in the change of fasting blood glucose in mmol/L between the intervention and control group
Change of lipids profiles | 6-month
  Difference in the change of lipids profiles (TC, HDL-C, LDL-C, TG) in mmol/L between the intervention and control group
Change of lipids profiles | 12-month
  Difference in the change of lipids profiles (TC, HDL-C, LDL-C, TG) in mmol/L between the intervention and control group
Change of lipids profiles | 3-month
  Difference in the change of lipids profiles (TC, HDL-C, LDL-C, TG) in mmol/L between the intervention and control group
Change of echocardiography parameters (IVSd、IVSs、LVPWd, LVPWs, LVEDD) | 6-month
  Difference in the change of echocardiography parameters (IVSd、IVSs、LVPWd, LVPWs, LVEDD, in millimetre[mm]) between the intervention and control group
Change of echocardiography parameters (IVSd、IVSs、LVPWd, LVPWs, LVEDD) | 12-month
  Difference in the change of echocardiography parameters (IVSd、IVSs、LVPWd, LVPWs, LVEDD, in millimetre[mm]) between the intervention and control group
Change of echocardiography parameters (IVSd、IVSs、LVPWd, LVPWs, LVEDD) | 3-month
  Difference in the change of echocardiography parameters (IVSd、IVSs、LVPWd, LVPWs, LVEDD, in millimetre[mm]) between the intervention and control group
Change of 24-h urine microalbumin | 6-month
  Difference in the change of 24-h urine microalbumin (mg/L) between the intervention and control group
Change of 24-h urine microalbumin | 12-month
  Difference in the change of 24-h urine microalbumin (mg/L) between the intervention and control group
Change of 24-h urine microalbumin | 3-month
  Difference in the change of 24-h urine microalbumin (mg/L) between the intervention and control group
Change of 24-h urine creatinine | 6-month
  Difference in the change of 24-h urine creatinine (umol/L) between the intervention and control group
Change of 24-h urine creatinine | 12-month
  Difference in the change of 24-h urine creatinine (umol/L) between the intervention and control group
Change of 24-h urine creatinine | 3-month
  Difference in the change of 24-h urine creatinine (umol/L) between the intervention and control group
Change of echocardiography parameters (LVEF) | 6-month
  Change of echocardiography parameters (LVEF)
Change of echocardiography parameters (LVEF) | 12-month
  Change of echocardiography parameters (LVEF)
Change of echocardiography parameters (LVEF) | 3-month
  Change of echocardiography parameters (LVEF)
Change of carotid intima-media thickness | 6-month
  Difference in the change of carotid intima-media thickness(CIMT) assessed by carotid ultrasound between the intervention and control group
Change of carotid intima-media thickness | 12-month
  Difference in the change of carotid intima-media thickness(CIMT) assessed by carotid ultrasound between the intervention and control group
Change of carotid intima-media thickness | 3-month
  Difference in the change of carotid intima-media thickness(CIMT) assessed by carotid ultrasound between the intervention and control group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang X, Luo T, Yang Y, Zhou Y, Hou J, Wang P. Unilateral chemical ablation of the adrenal gland lowers blood pressure and alleviates target organ damage in spontaneously hypertensive rats. Hypertens Res. 2023 Dec;46(12):2693-2704. doi: 10.1038/s41440-023-01444-2. Epub 2023 Oct 3. PMID 37789113
- [Background] Zhou Y, Wang X, Hou J, Wan J, Yang Y, Liu S, Luo T, Liu Q, Xue Q, Wang P. A controlled trial of percutaneous adrenal arterial embolization for hypertension in patients with idiopathic hyperaldosteronism. Hypertens Res. 2024 Feb;47(2):311-321. doi: 10.1038/s41440-023-01420-w. Epub 2023 Aug 29. PMID 37644179
- [Background] Zhou Y, Wang D, Liu Q, Hou J, Wang P. Case report: Percutaneous adrenal arterial embolization cures resistant hypertension. Front Cardiovasc Med. 2022 Oct 11;9:1013426. doi: 10.3389/fcvm.2022.1013426. eCollection 2022. PMID 36304542
- [Background] Zhou Y, Liu Q, Wang X, Wan J, Liu S, Luo T, He P, Hou J, Pu J, Wang D, Liang D, Yang Y, Wang P. Adrenal Ablation Versus Mineralocorticoid Receptor Antagonism for the Treatment of Primary Aldosteronism: A Single-Center Prospective Cohort Study. Am J Hypertens. 2022 Dec 8;35(12):1014-1023. doi: 10.1093/ajh/hpac105. PMID 36205513